CLINICAL TRIAL: NCT00998907
Title: Pathway Driven Study to Evaluate the Incidence of Wound Infections and Incisional Hernias After Laparotomy and Fascial Closure With PDS*Plus Sutures
Brief Title: PDS*Plus and Wound Infections After Laparotomy
Acronym: PDS*plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Principal Investigator, Christoph Justinger, Priciple Investigator, University Hospital, Saarland
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/2009
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Wound Infection; Incisional Hernia
Keywords: Open Abdominal Surgery; Fascial Closure
MeSH Terms: conditions — Wound Infection; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDS II (Active Comparator): PDS II® loop suture is used for abdominal wall closure
  Interventions: Device: PDS II
- PDS plus (Experimental): antibacterial coated "PDS plus" is used for abdominal wall closure
  Interventions: Device: PDS plus

INTERVENTIONS:
Device: PDS plus — triclosan-coated polydiaxanon 910 suture materials with antiseptic activity (PDS plus®, Ethicon GmbH, Norderstedt, Germany)
  Other Names: PDS plus®
  Arms: PDS plus
Device: PDS II — polyglactin 910 suture material for abdominal wall closure
  Arms: PDS II

SUMMARY:
The aim of this study is to ascertain if the use of PDS plus® reduces the number of wound infections and incisional hernia after midline and transverse laparotomy comparing to polyglactin suture.

DETAILED DESCRIPTION:
All patients are treated using clinical pathways (CP) to standardise surgical procedures in our high volume centre. Part of the clinical process management was the standardisation of wound incision and abdominal wall closure.

Wound closure is achieved using continuous absorbable loop suture. The suture length to incision length ratio is at least 4:1. The running sutures are 1 cm apart and at least 1.5 cm from the wound edge. In the first time period , the CP step for fascia closure foresees a triclosan-coated PDS 910 loop suture (PDS plus®, Ethicon GmbH, Norderstedt, Germany). In the second time period the CP step will be altered to the use of PDS loop suture (PDS II®, Ethicon GmbH, Norderstedt, Germany). The CP- step is changed every 100 patients to cluster-randomize the patients. The primary outcome is the number of wound infections. Together with this the number of incisional hernia will be recorded. Patients demographic and disease as well as procedure related data are collected in a clinical information system (ISHmed on SAP platform, GSD, Berlin, Germany) prospectively. Risk factors for poor wound healing, such as operation time, patients age, sex, body mass index, blood loss, peritonitis, antibiotics, and performance level classified according to the American Society of Anesthesiologists (ASA), are collected prospectively to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* surgical pathologies accessed via midline or transverse abdominal incision
* primary fascial closure

Exclusion Criteria:

* pregnancy
* age under 18 years
* open abdominal treatment
* known hypersensitivity against PDS/Triclosan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1042 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The number of wound infections | 30 days after the operation

SECONDARY OUTCOMES:
The number of incisional hernias. | 6 month
The number of incisional hernia- long time follow up | 12 month
  number of incisional hernia after 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Justinger, M.D., Principal Investigator — Department of General, Visceral, Vascular and Pediatric Surgery, University of Saarland, D-66421 Homburg/Saar, Germany; Martin K Schilling, M.D., FRCS, Study Director — Department of General, Visceral, Vascular and Pediatric Surgery, University of Saarland, D-66421 Homburg/Saar, Germany
Locations (1):
- Department of General, Visceral, Vascular and Pediatric Surgery, University of Saarland,, Homburg/Saar, Germany

REFERENCES:
- [Background] Justinger C, Moussavian MR, Schlueter C, Kopp B, Kollmar O, Schilling MK. Antibacterial [corrected] coating of abdominal closure sutures and wound infection. Surgery. 2009 Mar;145(3):330-4. doi: 10.1016/j.surg.2008.11.007. Epub 2009 Jan 25. PMID 19231586
- [Derived] Justinger C, Slotta JE, Ningel S, Graber S, Kollmar O, Schilling MK. Surgical-site infection after abdominal wall closure with triclosan-impregnated polydioxanone sutures: results of a randomized clinical pathway facilitated trial (NCT00998907). Surgery. 2013 Sep;154(3):589-95. doi: 10.1016/j.surg.2013.04.011. Epub 2013 Jul 13. PMID 23859304
- See also: Dept. of General Surgery, Visceral, Vascular and Pediatric Surgery, University Hospital of Saarland — http://www.uniklinikum-saarland.de/de/einrichtungen/kliniken-und-institute/chirurgie/allgemeinchirurgie